CLINICAL TRIAL: NCT05331157
Title: Ultrasonically Versus Conventional Palpation for Epidural Analgesia in Pediatrics Undergoing Midabdominal Urological Operations
Brief Title: Ultrasound Epidural Technique
Acronym: US_epidural
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, Assistant Professor of Anesthesia and Surgical Intensive Care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ultrasound epidural
Record Dates: First submitted 2022-03-28; First posted 2022-04-15 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Pediatric- Epidural Analgesia -Palpation-ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patients will be randomly assigned to 2 equal groups (ultrasonography and palpation; 55 subjects in each group) using the permuted block randomization method with randomly selected block sizes of 4 and 6. The group allocation codes were concealed in sequentially numbered, opaque, sealed envelopes that were opened only after assessing the eligibility and obtaining the consent from the parents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- palpation group (No Intervention): In lateral decubitus position, the conventional palpation technique will be used to detect the epidural space. The midline will be identified by palpation of the spinous processes. Through the Tuffier's line, L5 spine then, the two intervertebral spaces (L3-4 and L2-3) will be detected and the middle of each intervertebral space will be marked with selection of the widest space.
  After sterilization of the patient's skin the needle will be inserted to detect the epidural space by using loss of resistance to saline
- Ultrasonography group (Experimental): In lateral decubitus position, a curved array probe will be utilized to scan the sacrum in the longitudinal paramedian plane, then the probe will be moved upwards to detect the L5-S1, L4-5, L3-4 and L2-3 intervertebral spaces then turned 90º to the transverse plane and used to scan L3-4 and L2-3 spaces inside the 2 spaces, midline will be detected by noting the site of spinous processes with selection of the space with the best sonographic image quality. Then skin surface at the middle of the long and short axis of the probe will be marked horizontally. If the 2 spaces have the same image quality, L2-3 space will be chosen for the entrance of epidural needle. After sterilization of the patient's skin the needle will be inserted to detect the epidural space by using loss of resistance to saline
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — the efficacy of prepuncture ultrasonography to facilitate epidural block in pediatric patients undergoing elective urological operations compared with the conventional anatomical landmark technique
  Arms: Ultrasonography group

SUMMARY:
Epidural analgesia for abdominal surgeries provides numerous advantages for both neonates and children. The anatomical identification of the intervertebral space to access the epidural space is not constantly easy this is due uncertainty of the direction of the needle angle and the difficulty to estimate the epidural depth in spite of the skill of the operator. This can lead to more puncture attempts, inducing more pain or discomfort and even failure of epidural access.

Pre-procedure neuraxial ultrasound (US) imaging facilities the identification of the chosen intervertebral space, the depth of the epidural space and so the selection of best point and angle for the needle insertion

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of prepuncture ultrasonography to facilitate epidural block in pediatric patients undergoing elective urological operations compared with the conventional anatomical landmark technique

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged from 1 to 12 years old
* Both genders
* American Society of Anesthesiologists (ASA) physical status I,II, III
* Scheduled for open midabdominal urological surgeries under general anesthesia

Exclusion Criteria:

* Pediatric patients aged less than 1 or more than 12 years old
* American Society of Anesthesiologists (ASA) physical status Iv
* Parents' refusal to participate in the study
* Any contraindication to epidural block (as severe infection at the puncture site, coagulopathy or hemodynamically unstable patients)
* Neuromuscular diseases
* Severe spinal deformity
* History of allergy to the anesthetic drugs

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
the rate of a successful reaching to the epidural space from the first needle pass | minutes
  incidence after insertion of the epidural needle into the skin till reaching the epidural space

SECONDARY OUTCOMES:
the rate of a successful reaching to the epidural space from the first skin puncture | minutes
  incidence after insertion of the epidural needle into the skin till reaching the epidural space
The number of performed skin punctures by the epidural needle | minutes
  number after insertion of the epidural needle into the skin till reaching the epidural space
The number of needle passes from the same skin puncture required for reaching the epidural space | minutes
  number from the skin puncture done by the epidural needle till removing the epidural needle from this the skin puncture
The epidural space demarcation time by the ultrasound | minutes
  The time from placing the ultrasound probe on the skin until the skin marking is completed at L3-4 and L2-3 space
The epidural space demarcation time by the landmark | minutes
  The time from start skin palpation til the skin marking is completed at L3-4 and L2-3 space
The procedure time which is the time from the needle insertion into the skin until reaching the epidural space | minutes
Incidence of intraoperative hypertension (as increase in systolic blood pressure (SBP) by more than 20% from the basal) | allover the surgery (minutes)
  mmHg
Incidence of intraoperative tachycardia (as increase in heart rate by more than 20% from the basal) | allover the surgery (minutes)
  beat per minutes
The procedure time | minutes
  from the needle insertion into the skin till entering the epidural space
pain score using "face, leg, activity, cry, consolability" (FLACC) scale | 30 minutes after the patient has transferred to the recovery room
  five criteria, which are each assigned a score of 0, 1 or 2

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University-Emergency hospital-ICU, Al Mansurah, Egypt